CLINICAL TRIAL: NCT07068087
Title: Efficacy of Pre-operative Silodosin on Facilitating Insertion of Ureteral Access SheathPrior to Retrograde Intra Renal Surgery: A Randomized Controlled Study
Brief Title: Silodosin in Facilitating Flexible Uretroscopy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Younan Ramsis, Lecturer of urology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MS 766/2024
Record Dates: First submitted 2025-06-10; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Stone Ureter; Stone, Kidney
Keywords: Retrograde Intra Renal Surgery (RIRS); Flexible uretroscopy; Laser disintegration; Alpha blocker selective; Silodosin
MeSH Terms: conditions — Ureterolithiasis; Kidney Calculi | interventions — silodosin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receiving Sioldosin 8 mg prior to intervention (Active Comparator)
  Interventions: Procedure: Preoperative sioldosin to facilitate ureteric access sheath insertion in RIRS
- Receiving Placebo prior to intervention (Placebo Comparator)
  Interventions: Procedure: ureteric access sheath insertion in RIRS without silodosin (Placebo)

INTERVENTIONS:
Procedure: Preoperative sioldosin to facilitate ureteric access sheath insertion in RIRS — group A (study group) that included 21 patients who received silodosin 'one capsule 8 mg per day for 1 week preoperatively
  Arms: Receiving Sioldosin 8 mg prior to intervention
Procedure: ureteric access sheath insertion in RIRS without silodosin (Placebo) — group B (study group) that included 21 patients who received Placebo'one capsule per day for 1 week preoperatively
  Arms: Receiving Placebo prior to intervention

SUMMARY:
This study aims to provide robust evidence on whether a specific, potent pre-operative medication (silodosin) can make the critical step of ureteral access (UAS placement after dilation) easier and safer during f-URS for kidney stones in non-stented patients, potentially reducing complications and the need for pre-stenting.

DETAILED DESCRIPTION:
This study specifically evaluates the effect of administering pre-operative silodosin (8mg daily for one week) on facilitating ureteral dilation prior to ureteral access sheath (UAS) placement during flexible ureteroscopy (f-URS), aiming to leverage the drug's potent ureteral smooth muscle relaxation to ease mechanical dilation with Teflon dilators (6-14Fr) and subsequent UAS insertion. Its primary endpoint directly measures the ease of UAS placement (categorized as smooth, resistant, or failed) after sequential dilation. To objectively assess safety, post-operative diagnostic ureteroscopy by a second surgeon grades ureteral wall injuries using a specific 5-grade scale. Employing a rigorous randomized, placebo-controlled trial (RCT) design with strict criteria (non-stented patients, stone burden 1-2 cm, no prior interventions), the study also evaluates secondary outcomes including ureteral injury severity, stone-free rates (SFR), post-operative pain (VAS), complications, hospital stay length, and medication side effects.

ELIGIBILITY:
Inclusion Criteria:

* adult male or female
* single renal or ureteric stone
* 1 to 2 cm in size.

Exclusion Criteria:

* pregnant women
* Untreated urinary tract infections
* Uncorrected bleeding disorders or coagulopathies
* Bilateral ureteric stones or multiple ipsilateral ureteric stones
* ureteral stricture,
* Patients who had previous ureteric stenting

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Assess success of ureteric access sheath placement. | during the operation in the OR
  assess success of ureteric access sheath placement as follows: 1. spontaneous passage of UAS without dilatation or 2. passage of UAS after dilatation or 3. failure of the UAS insertion.

SECONDARY OUTCOMES:
Operative time | from time of induction of anaesthesia in surgery till the end of procedure.
Cost of the procedure | from admission and through study completion
  Overall cost of each procedure included cost of standard procedure of flexible URS added to cost of medication prior to operations. If any case needed ureteral dilatation, the cost of dilators was added. Also, in case of complications occurred, additional cost of management of these complications was added. Finally, in cases of failed UAS insertion, the cost of auxiliary procedure was added. Cost was calculated initially in Egyptian pounds and was converted to U.S dollars for standardization.
complications | Perioperative and up to 24 weeks
  Assess postoperativePain, fever and Residual stones

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud A. Mohammed, M.D., Study Chair — Ain Shams University; Younan R. Samir, M.D., Study Director — Ain Shams University
Locations (1):
- Ain Shams University hospitals (Demerdash), Cairo, Abasia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benedict, A., Rajenthiran, V., & Eswaramurthy, A. (2021). Effects of silodosin, darifenacin, and combination therapy for the treatment of ureteral stent related discomforts. International Surgery Journal, 8(10), 3031-3035.
- [Background] Alsaikhan B, Koziarz A, Lee JY, Pace KT. Preoperative Alpha-Blockers for Ureteroscopy for Ureteral Stones: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Endourol. 2020 Jan;34(1):33-41. doi: 10.1089/end.2019.0520. Epub 2019 Oct 9. PMID 31507224
- [Background] Alaridy, H. M., Zwain, K. M. A., Al-Mosawi, H. Q., & Hadi, N. R. (2020). Comparison of silodosin, tadalafil and combinations prior to ureteroscopic management of ureteral stones. Systematic Reviews in Pharmacy, 11(4), 238-242.